CLINICAL TRIAL: NCT02189395
Title: Comparison of Neutral Protamine Hagedorn (NPH) and Lantus Based Insulin Regimen in the Management of Hypoglycemia in the Hospitalized Patients in Noncritical Care Setting
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty in subject recruitment
Sponsor: Riverside University Health System Medical Center (Other)
Responsible Party: Principal Investigator, Iqbal Munir, MD, PhD, Principal Investigator, Riverside University Health System Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 437860
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; Uncontrolled blood glucose; insulin; glargine; NPH
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NPH and regular insuline group (Experimental): For the group receiving NPH and regular 2/3 and 1/3 formula will be followed. If Nil per os (NPO), patient will receive NPH twice daily but AM dose will equal to PM dose. Regular insulin given along with NPH will be held while patient is NPO. A correctional dose of regular insulin will be given for any blood glucose >180 mg/dL. If subjects were not eating, they could also receive correctional doses of regular insulin. Correctional insulin could be given four times daily with meals or at bedtime.
  Interventions: Drug: NPH and regular insulin
- glargine and humalog group (Active Comparator): Half of the total insulin dose will be given as glargine once daily, either in the AM or in the PM, depending on when the patient was enrolled. The other half of the total daily insulin dose was given as humalog; doses were divided equally between breakfast, lunch, and dinner. An additional correctional dose of humalog will be given for any blood glucose >180 mg/dL. If subjects were not eating, they received glargine once daily and could also receive correctional doses of humalog. Correctional humalog could be given four times daily with meals or at bedtime.
  Interventions: Drug: glargine and humalog

INTERVENTIONS:
Drug: NPH and regular insulin
  Arms: NPH and regular insuline group
Drug: glargine and humalog
  Arms: glargine and humalog group

SUMMARY:
The goal of the current study is to determine difference in glycemic control between traditional split mix regimen with Neutral Protamine Hagedorn (NPH) and regular insulin vs basal bolus regimen with glargine and humalog in a population of type 2 diabetes commonly encountered in the investigators county hospital setting which include newly diagnosed type 2 patients and patients on relatively high dose of insulin (dose >0.4 units/kg body weight. Primary outcome of the study is to determine differences in glycemic control between treatment group as measured by the mean daily blood glucose. Secondary outcome is to measure number of hypoglycemic events, number of severe hypoglycemia and length of hospital stay.

DETAILED DESCRIPTION:
The effect of insulin depends not only on the pharmacokinetics and pharmacodynamics of a particular preparation, but also on patient specific factors which includes state of inflammation, obesity etc. Although effect on glucose disposal is the central to insulin action, there could be differences of insulin action on other metabolic parameters. It is not known if there is a difference in suppression of inflammation with improved glycemic control which could vary with analog insulin. It is unknown if natural insulin (NPH, recombinant human insulin with protamine) differs from insulin analogs (glargine and detemir, made by substituting amino acid in the native sequence) in terms of metabolic outcome other than glucose disposal.

At this point it is uncertain if there is any clear benefit of use of lantus over NPH in inpatient glycemic management. Currently, both lantus and NPH based regimen is practiced in inpatient hospital setting. Current practice of inpatient insulin regimen is based more on familiarity of physicians with a particular insulin type and personal preference rather than evidenced based knowledge. Lantus is an expensive insulin preparation compared to NPH with uncertain benefit in inpatient setting. Current research proposal will compare this two insulin based regimen in the management of diabetes of hospitalized patients. Information obtained through this research will guide the investigators practice in this institution as well as in other institutions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type II diabetes regardless of duration of diagnosis with an admission blood glucose level between 140 mg/dL to 400 mg/dL will be included in the study.
* Other inclusion criteria are as follows:

  * age 18-80 years old
  * treated with diet alone
  * any combination of oral anti-diabetic agents or insulin treatment with any dosage before admission.

Exclusion Criteria:

* Hyperglycemia without a known history of diabetes
* H/o recent cardiac surgery (within 6 months)
* Impaired renal function (glomerular filtration rate less than 45)
* History of diabetic ketoacidosis
* Diabetes mellitus type 1
* Pregnancy
* Patients on steroid treatment
* Known hypopituitarism or adrenal insufficiency
* Known hypoglycemia of unawareness
* Length of stay <48 h
* And severe liver disease and patent admitted in intensive care unit.
* Patients already received an insulin dose greater than 0.5 units/kg body weight after admission prior to initiation of study protocol will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
difference in glycemic control between treatment groups as measured by the mean daily blood glucose | Duration of hospital stay, up to 24 weeks
  Primary outcome of the study is to determine differences in glycemic control between treatment group as measured by the mean daily blood glucose

SECONDARY OUTCOMES:
number of hypoglycemic events | duration of hospital stay, up to 24 weeks
  number of hypoglycemic events

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside County Regional Medical Center, Moreno Valley, California, United States